CLINICAL TRIAL: NCT04801381
Title: WATER III: Aquablation vs. Transurethral Laser Enucleation of Large Prostates (80-180ml) in Benign Prostatic Hyperplasia
Brief Title: WATER III: Aquablation vs. Transurethral Laser Enucleation of Large Prostates (80 - 180mL) in Benign Prostatic Hyperplasia
Acronym: WATER III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: PROCEPT BioRobotics (Industry)
Responsible Party: Principal Investigator, Manuel Ritter, Univ.-Prof. Dr. med. Manuel Ritter, University of Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-202001
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: BPH With Urinary Obstruction With Other Lower Urinary Tract Symptoms
Keywords: Aquablation therapy; Laserenucleation; HoLEP; ThuLEP

STUDY DESIGN:
Intervention Model Description: randomized and non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquablation therapy (Active Comparator): Aquablation therapy: Computer-assisted transurethral ablation of prostate tissue using a high-pressure water jet. Subsequent removal of residual ablated tissue at the bladder neck and haemostasis by transurethral electroresection (TUR).
  Interventions: Procedure: Aquablation therapy
- Transurethral laser enucleation (Active Comparator): Transurethral laser enucleation of the prostate using thulium laser (ThuLEP) or holmium laser (HoLEP).
  Interventions: Procedure: Transurethral laser enucleation

INTERVENTIONS:
Procedure: Aquablation therapy — Aquablation is carried out with the AQUABEAM Robotic System®, PROCEPT BioRobotics, Redwood City, CA, USA
  Arms: Aquablation therapy
Procedure: Transurethral laser enucleation — Transurethral laser enucleation is performed according to the standard established at the respective test center. Included laser techniques: Holmium laser (HoLEP) and Thulium laser (ThuLEP).
  Arms: Transurethral laser enucleation

SUMMARY:
Comparative analysis of efficacy and safety of Aquablation (AQUABEAM Robotic System®, PROCEPT BioRobotics, Redwood City, CA, USA) and transurethral laser enucleation as surgical therapy for benign prostatic hyperplasia with large prostates (80-180ml).

DETAILED DESCRIPTION:
Prospective randomized and non-randomized cohort, two-arm multicenter trial two arm multicenter trial to evaluate the efficacy and safety of Aquablation (AQUABEAM Robotic System®, PROCEPT BioRobotics, Redwood City, CA, USA) compared to transurethral laser enucleation - the current reference standard of minimal invasive therapy for benign prostatic hyperplasia in large prostates (80-180ml).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45 - 80 years
2. International Prostate Symptom Score (IPSS) ≥ 8
3. Prostate size (measurement by transrectal ultrasound): 80 - 180 mL
4. Subject has diagnosis of LUTS (Lower urinary tract symptoms) due to BPH (Benign Prostatic Hyperplasia)
5. Patient is mentally capable and willing to sign a study-specific consent form
6. Subjects with the ability to follow study instructions and likely to attend and complete all required visits
7. Written informed consent

Exclusion Criteria:

1. Body mass index ≥ 42
2. Suspected or history of prostate cancer
3. Suspected or history of bladder cancer
4. Bladder stone
5. Indwelling catheter for more than 3 months before baseline
6. Active urinary tract infection
7. History of urethral stricture or bladder neck stenosis
8. Damage of the external urethral sphincter
9. Previous prostate surgery or history of lower urinary tract surgery (e.g. urinary diversion, artificial sphincter or penile prosthesis)
10. Use of anticoagulants (if medication cannot be stopped before and after procedure) or known coagulopathy (except ASS 100mg/d).
11. Contraindications for general and spinal anaesthesia
12. The investigator considers a pre-existing condition or the subject's life circumstances to be problematic for the conduct of the study and the completion of the follow-up investigations
13. Subject is unwilling to accept a blood transfusion if required
14. Subject is not able to give consent
15. Subject without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial
16. Simultaneously participation in another clinical trial in the field of urology
17. Known or persistent abuse of medication, drugs or alcohol

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 202 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 3 months after index procedure
  Primary efficacy endpoint is defined as IPSS (International Prostate Symptom Score) change
Primary Safety Endpoint | Through 3 months after index procedure
  Primary safety endpoint is defined as the occurrence of an Adverse Event rated by the investigator as related or unrelated to the study procedure, classified as Clavien Dindo grade 2 or higher or any grade 1 event resulting in persistent disability, such as ejaculatory or erectile dysfunction or incontinence, as evidenced through 3 months after treatment.

SECONDARY OUTCOMES:
Change in IPSS | 1,6,12,24,36,48 and 60 months after index procedure
  Change in IPSS (International Prostate Symptom Score)
Change in IIEF 5/SHIM | 3,6,12,24,36,48 and 60 months after index procedure
  Change in IIEF5/SHIM (International Index of Erectile Function)
Change in MSHQ-EjD-SF | 3,6,12,24,36,48 and 60 months after index procedure
  Change in MSHQ-EjD-SF (Male Sexual Health Questionnaire for Ejaculatory Dysfunction Short Form)
Change in Dysuria Questionnaire | 1,3,6,12,24,36,48 and 60 months after index procedure
  Change in Dysuria Questionnaire
Change in ICIQ-UI-SF | 1,3,6,12, 24,36,48 and 60 months after index procedure
  Change in ICIQ-UI-SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form)
Post void residual urine | day 2-5, 3 months, 6 months, 12 months and 36 months after index procedure
  Reduction of Post void residual urine
Qmax, Uroflowmetry | day 2-5, 3 months, 6 months, 12 months and 36 months after index procedure
  Changes of maximum flow rate (Qmax) measured by Uroflowmetry
Prostate volume reduction | comparison of Visit 5 (3 months) and visit 1 (baseline)
  Prostate volume reduction
Number of re-interventions | Through 60 months after index procedure
  Number of re-interventions defined as need for additional tissue resection following the index procedure due to BPH.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ritter, Univ.-Prof. Dr. med., Principal Investigator — Department of Urology, University of Bonn
Locations (5):
- Germany (3):
  - Department of Urology, University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Department of Urology, Augusta-Kranken-Anstalt, Bochum Mitte, Bochum, North Rhine-Westphalia
  - Department of Urology, University Hospital Bonn, Bonn, North Rhine-Westphalia
- United Kingdom (2):
  - Frimley Health NHS Foundation Trust, London
  - Guy's and St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No